CLINICAL TRIAL: NCT06932003
Title: A Phase Ic/II Clinical Study to Explore the Safety, Tolerability, Efficacy, and Pharmacokinetics of Multiple Oral Doses of LT-002-158 Tablets in Chinese Adult Patients With Hidradenitis Suppurativa
Brief Title: A Study to Explore the Safety, Tolerability, Efficacy, and Pharmacokinetics of LT-002-158 Tablets in Chinese Adult Patients With Hidradenitis Suppurativa
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leadingtac Pharmaceutical (Shaoxing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT2158CHN005
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LT-002-158 Tablets (Experimental)
  Interventions: Drug: LT-002-158 Tablets

INTERVENTIONS:
Drug: LT-002-158 Tablets — The subjects will orally administered LT-002-158 tablets once a day.

SUMMARY:
This study is a Phase Ic/II clinical trial conducted in Chinese patients with moderate-to-severe hidradenitis suppurativa (HS), aiming to evaluate the safety and efficacy of LT-002-158 tablets in the treatment of moderate-to-severe HS.

The study consists of two parts. The Phase Ic portion employs an open-label, single-arm design to primarily investigate the safety and tolerability of LT-002-158 tablets in patients with moderate-to-severe HS. The Phase II study adopts a randomized, double-blind, placebo-controlled, parallel-group design, with an open-label, single-arm extension phase, to primarily assess the therapeutic efficacy of LT-002-158 tablets in patients with moderate-to-severe HS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years (inclusive), with body mass index (BMI) between 17.5 and 40.0 kg/m² (inclusive) and body weight ≥45.0 kg;
2. Diagnosis of hidradenitis suppurativa (HS) with disease duration of at least 6 months prior to enrollment;
3. Have inadequate response or intolerance to prior HS treatments and are suitable candidates for this study on investigator's judgment;
4. Total count of abscesses and inflammatory nodules ≥4 at baseline;
5. No pregnancy plans during the study and for 6 months after the last dose, with agreement to use effective contraception methods;
6. Understand and voluntarily sign the informed consent form; Willing and able to to complete patient diary entries as required by the protocol;
7. The subject is willing and able to comply with all protocol requirements by investigator's judgment.

Exclusion Criteria:

1. Presence of >20 fistulas or deeply extensive coalescing lesions;
2. Other significant dermatological conditions that may interfere with efficacy evaluation or require concomitant treatment (e.g., seborrheic dermatitis), or any skin conditions deemed by investigators as potentially affecting study assessments (e.g., tattoos, scars);
3. Any of the following comorbidities:

   1. Active tuberculosis;
   2. Active hepatitis B/C, syphilis, or human immunodeficiency virus (HIV) infection;
   3. Severe cardiovascular diseases including: Congestive heart failure (NYHA class ≥II); Angina pectoris >grade 1; Known structural heart disease; Major cardiovascular events within screening period (myocardial infarction, unstable angina, acute coronary syndrome, stroke or transient ischemic attack, etc.); Ventricular fibrillation; TDP; atrial fibrillation; Unexplained syncope of non-cardiac origin;
   4. Immunodeficiency or immune-related disorders (organ/bone marrow transplantation, splenectomy, IgG4-related disease, vasculitis, etc.) or active autoimmune diseases requiring treatment (psoriasis, atopic dermatitis, rheumatoid arthritis, etc.);
   5. History or symptoms of malignancy in any organ system within 5 years prior to screening, regardless of treatment status or evidence of recurrence/metastasis (except appropriately treated non-metastatic cutaneous carcinoma in situ or cervical basal/squamous cell carcinoma in situ);
   6. Gastrointestinal disorders or surgeries (gastrectomy, gastric bypass, etc.) that may affect oral drug absorption;
4. Family history of sudden death or long QT syndrome, or personal history of congenital/medication-induced long QT syndrome;
5. Any of the following laboratory abnormalities:

   1. Estimated glomerular filtration rate (eGFR) or creatinine clearance (CrCl) <60 mL/min/1.73m²;
   2. Total bilirubin ≥1.5×upper limit of normal (ULN);
   3. ALT ≥1.5×ULN or AST ≥1.5×ULN;
   4. Hemoglobin <9.0 g/dL, WBC <3.0×10⁹/L, neutrophils <1.5×10⁹/L, lymphocytes <0.75×10⁹/L, platelets <100×10⁹/L;
   5. Serum potassium, magnesium, or calcium below lower limit of normal;
   6. QTcF >450 ms or QRS >110 ms on screening ECG;
   7. Blood pressure ≥150/90 mmHg despite antihypertensive treatment;
6. Use of adalimumab or other biologics within 8 weeks or 5 half-lives prior to first dose (whichever longer) (≤20% of enrolled subjects may have prior biologic exposure without treatment failure);
7. Systemic antibiotic therapy within 2 weeks or systemic retinoid therapy within 4 weeks prior to first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events | Day 1-Day 42
  Including adverse events (TEAEs) and serious adverse events that occurred during the study period; Clinically significant changes observed in laboratory tests, 12 lead electrocardiograms, vital signs, and physical examinations during the study period.

SECONDARY OUTCOMES:
Area under the curve plasma concentration from time zero to last measurable concentration [AUC(0-last)] | Day 1-Day 42
Maximum observed plasma concentration (Cmax) | up to 42 days
Time to maximum observed plasma concentration (Tmax) | up to 42 days